CLINICAL TRIAL: NCT04761133
Title: Antiseptic Pleural Irrigation for Patients With Pleural Infection
Brief Title: Antiseptic Irrigation for Pleural Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Maged Hassan, Clinical Lecturer, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04/24/11/10/2020
Record Dates: First submitted 2021-02-13; First posted 2021-02-18 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Pleural Infection
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pleural irrigation with antiseptic (Experimental): Two applications of 100-250 ml solution of 2% povidone-iodine will be irrigated into the pleural space of eligible patients 12 hours apart. The tube will be clamped for 15 minutes after irrigation and the patient will be asked to change position frequently during this period. The first dose will be applied 24-72 hours after tube insertion.
  Interventions: Drug: Povidone-Iodine pleural irrigation
- No pleural irrigation (No Intervention): Standard care

INTERVENTIONS:
Drug: Povidone-Iodine pleural irrigation — Irrigation of the infected pleural cavity with an antiseptic solution to reduce microbial load
  Other Names: Betadine
  Arms: Pleural irrigation with antiseptic

SUMMARY:
The antiseptic povidone-iodine can safely be instilled into the pleural for the purpose of pleurodesis. Pleural irrigation with antiseptics is used in adults with open drainage for chronic empyema and has been described in the acute management of paediatric pleural infection.

This study will investigate the safety and usefulness of povidone-iodine pleural irrigation in 15 eligible patients recruited to the Pleural Infection Cohort Study (PICS) with acute pleural infection. A matched control group will be used and will be composed of 15 patients previously recruited to PICS without receiving povidone-iodine pleural irrigation.

DETAILED DESCRIPTION:
Pleural infection is a condition that requires hospitalization for management and is associated with significant in-hospital morbidity and mortality. Predictors of poor outcome include advancing age, poor nutrition, hospital-acquired infection and impaired renal function. Medical management is centred on appropriate antibiotic treatment and fluid drainage usually by the means of an intercostal tube. Up to 30% of patients fail medical treatment and referred for surgery. A recent systematic review of adults patient with pleural infection has shown that the demographics of patients with pleural infection are different in patients from high-income vs lower income countries; the latter being of younger age and lower comorbidity burden. However, the results of the review did not show significant differences in patient outcomes. The same systematic review pointed to the need for more data from patients residing in lower income countries given that the majority of data is contributed by studies from higher income countries.

This platform study aims to prospectively investigate the incidence of pleural infection in a large tertiary centre gathering demographic and clinical data about patients recruited. In addition, the study will examine the different treatment offered and how this related to in-hospital outcomes (length of hospital stay, rate of referral to surgery and mortality).

The study will be designed as a modified trial within cohort (TwiC) study. PICS will primarily aim to recruit patients prospectively to gather clinical and demographic data on patients admitted with pleural infection in addition to clinical data on tests performed and treatments received as part of the standard care. The in-patient outcomes will be recorded at the time of discharge data or death, whichever is earlier. Within the TWIC design, PICS will be a platform for recruiting patients to interventional trials for eligible patients within the cohort. As a planned sub-study, pleural antiseptics will be trialed within a subset of patients enrolled.

The antiseptic povidone-iodine can safely be instilled into the pleural for the purpose of pleurodesis. Pleural irrigation with antiseptics is used in adults with open drainage for chronic empyema and has been described in the acute management of paediatric pleural infection.

This sub-study will investigate the safety and usefulness of povidone-iodine pleural irrigation in 15 eligible adult patients recruited to PICS with acute pleural infection. A matched control group will be used and will be composed of 15 patients previously recruited to PICS without receiving povidone-iodine pleural irrigation.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to hospital with pleural infection and had a chest tube inserted for treatment of the infection. Pleural infection will be defined by the presence of one of the following: a) the presence of pus in the pleural space; b) positive pleural fluid gram stain or culture; or c) pleural fluid pH < 7.2 or pleural fluid glucose < 40 mg/dL in the setting of acute respiratory infection.
* Pleural collection is unilocular on pre-drainage imaging. Presence of septations on ultrasound examination is allowed.

Exclusion Criteria:

* Known or suspected thyroid disease
* Allergy to iodine
* Persistent large collection on follow up imaging 24-48 of post tube insertion that requires another drainage procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Within 24 hours after the second application of the study medication
  Number of subjects with any adverse event (new chest pain, fever, dyspnoea or oxygen desaturation)
Time to chest tube removal | Up to 8 weeks
  Number of days from tube insertion to tube removal

SECONDARY OUTCOMES:
Time to defervescence | Up to 8 weeks
  Numbers of days until resolution of fever
Length of hospital stay | Up to 8 weeks
  Number of days from admission/diagnosis until discharge from hospital
Incidence of need for additional aspiration/tubes | Up to 8 weeks
  Number of patients requiring additional drainage procedures during hospital admission
Incidence of medical treatment of failure | Up to 8 weeks
  Number of patients requiring surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maged Hassan, PhD, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
At completion of study assessments for the last recruited patients, data will be transferred from paper to electronic forms (spreadsheets) to allow statistical analysis. These spreadsheets will be stored securely after trial conclusion with the principal investigator and will be accessible to other members of the study team. Request to access study data by other teams will be expected via email and access will be granted by the principal investigator if the request is deemed reasonable.
Time Frame: From published to study results up until five years after study completion
Access Criteria: Access will be granted upon reasonable request via email to the principal investigator

REFERENCES:
- [Background] Davies HE, Davies RJ, Davies CW; BTS Pleural Disease Guideline Group. Management of pleural infection in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii41-53. doi: 10.1136/thx.2010.137000. No abstract available. PMID 20696693
- [Background] Corcoran JP, Psallidas I, Gerry S, Piccolo F, Koegelenberg CF, Saba T, Daneshvar C, Fairbairn I, Heinink R, West A, Stanton AE, Holme J, Kastelik JA, Steer H, Downer NJ, Haris M, Baker EH, Everett CF, Pepperell J, Bewick T, Yarmus L, Maldonado F, Khan B, Hart-Thomas A, Hands G, Warwick G, De Fonseka D, Hassan M, Munavvar M, Guhan A, Shahidi M, Pogson Z, Dowson L, Popowicz ND, Saba J, Ward NR, Hallifax RJ, Dobson M, Shaw R, Hedley EL, Sabia A, Robinson B, Collins GS, Davies HE, Yu LM, Miller RF, Maskell NA, Rahman NM. Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study. Eur Respir J. 2020 Nov 26;56(5):2000130. doi: 10.1183/13993003.00130-2020. Print 2020 Nov. PMID 32675200
- [Background] Maskell NA, Davies CW, Nunn AJ, Hedley EL, Gleeson FV, Miller R, Gabe R, Rees GL, Peto TE, Woodhead MA, Lane DJ, Darbyshire JH, Davies RJ; First Multicenter Intrapleural Sepsis Trial (MIST1) Group. U.K. Controlled trial of intrapleural streptokinase for pleural infection. N Engl J Med. 2005 Mar 3;352(9):865-74. doi: 10.1056/NEJMoa042473. PMID 15745977
- [Background] Cargill TN, Hassan M, Corcoran JP, Harriss E, Asciak R, Mercer RM, McCracken DJ, Bedawi EO, Rahman NM. A systematic review of comorbidities and outcomes of adult patients with pleural infection. Eur Respir J. 2019 Oct 1;54(3):1900541. doi: 10.1183/13993003.00541-2019. Print 2019 Sep. PMID 31391221
- [Background] Kim SY, Flory J, Relton C. Ethics and practice of Trials within Cohorts: An emerging pragmatic trial design. Clin Trials. 2018 Feb;15(1):9-16. doi: 10.1177/1740774517746620. Epub 2017 Dec 11. PMID 29224380
- [Background] Agarwal R, Khan A, Aggarwal AN, Gupta D. Efficacy & safety of iodopovidone pleurodesis: a systematic review & meta-analysis. Indian J Med Res. 2012 Mar;135(3):297-304. PMID 22561614
- [Background] Light RW. Parapneumonic effusions and empyema. Proc Am Thorac Soc. 2006;3(1):75-80. doi: 10.1513/pats.200510-113JH. PMID 16493154
- [Background] Togo S, Ouattara MA, Sangaré I, Saye J, Touré CAS, Maiga IB, et al. Management for Pediatric Pleural Empyema in Resource-Poor Country: Is Chest Tube Drainage with Antiseptic Lavage-Irrigation Better than Tube Thoracostomy Alone? SS 2015;06(12):541-8.

DOCUMENTS (1):
  • Study Protocol (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT04761133/Prot_000.pdf